CLINICAL TRIAL: NCT00788671
Title: A Phase II Study of the Levonorgestrel Intrauterine Device (Mirena) to Treat Complex Atypical Hyperplasia and Grade 1 Endometrioid Endometrial Carcinoma
Brief Title: Levonorgestrel-Releasing Intrauterine System in Treating Patients With Complex Atypical Hyperplasia or Grade I Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0094; NCI-2012-02118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0094 (Other: M D Anderson Cancer Center); P50CA098258 (NIH)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2022-04-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Atypical Endometrial Hyperplasia; Stage I Uterine Corpus Cancer AJCC v7; Stage IA Uterine Corpus Cancer AJCC v7; Stage IB Uterine Corpus Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (levonorgestrel-releasing intrauterine system) (Experimental): Patients undergo placement of a levonorgestrel-releasing intrauterine system.
  Interventions: Other: Laboratory Biomarker Analysis; Device: Levonorgestrel-Releasing Intrauterine System; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Levonorgestrel-Releasing Intrauterine System — Undergo placement of a levonorgestrel-releasing intrauterine system
  Other Names: Mirena
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well levonorgestrel-releasing intrauterine system works in treating patients with complex atypical hyperplasia or grade I endometrial cancer. High levels of estrogen can cause the growth of endometrial cancer cells. Progesterone can help balance the amount of estrogen present. Hormone therapy using levonorgestrel, a type of progesterone, may fight endometrial cancer by helping regulate hormone levels.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the levonorgestrel intrauterine device (IUD) (levonorgestrel-releasing intrauterine system) to treat complex atypical hyperplasia (CAH) and grade 1 endometrioid endometrial carcinoma (G1 EEC).

II. To determine if response to therapy can be predicted based on the molecular profile of the tumor or by change in gene expression after therapy.

SECONDARY OBJECTIVES:

I. To assess quality of life outcomes in patients treated with levonorgestrel IUD.

II. To document the toxicity profile of the levonorgestrel IUD in the treatment of complex atypical hyperplasia and grade 1 endometrioid endometrial cancer.

III. To evaluate the molecular profile of the hysterectomy specimen of patients treated with the levonorgestrel IUD. Compare molecular profile in pretreatment tissue to hysterectomy tissue between responders and non-responders to levonorgestrel IUD therapy.

IV. To evaluate long-term survival, disease status, and fertility outcomes in patients with levonorgestrel IUD.

OUTLINE:

Patients undergo placement of a levonorgestrel-releasing intrauterine system.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of complex atypical hyperplasia or endometrial biopsy within three months of study enrollment OR patients with a diagnosis of grade 1 endometrioid endometrial carcinoma on endometrial biopsy within three months of study enrollment in the presence of one or more of the following: 1)desire for future fertility 2)morbid obesity (body mass index > 40) 3)multiple co-morbidities (ASA Class 3 or 4)
* No prior treatment for diagnoses in inclusion criteria 1.
* Women of any racial or ethnic group.
* Ability to comply with endometrial biopsies every 3 months.
* Willing and able to sign informed consent.
* Age greater than 18 years.

Exclusion Criteria:

* Diagnosis of grade 1 endometrioid endometrial carcinoma without the presence of one of the 3 criteria mentioned in inclusion criteria 1.
* Diagnosis of grade 2 endometrioid endometrial carcinoma or higher on endometrial biopsy or on dilation and curettage specimen.
* Evidence of extrauterine spread of disease on imaging or during surgical evaluation.
* Congenital or acquired uterine anomaly which distorts the uterine cavity.
* Acute pelvic inflammatory disease.
* Acute liver disease or previously diagnosed liver tumor (benign or malignant).
* Conditions associated with increased susceptibility to infections with microorganisms. Such conditions include, but are not limited to, AIDS, leukemia and IV drug abuse.
* Genital actinomycosis.
* Current carcinoma of the breast.
* Current pregnancy.
* Breastfeeding mothers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-11-03 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2027-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Westin SN, Fellman B, Sun CC, Broaddus RR, Woodall ML, Pal N, Urbauer DL, Ramondetta LM, Schmeler KM, Soliman PT, Fleming ND, Burzawa JK, Nick AM, Milbourne AM, Yuan Y, Lu KH, Bodurka DC, Coleman RL, Yates MS. Prospective phase II trial of levonorgestrel intrauterine device: nonsurgical approach for complex atypical hyperplasia and early-stage endometrial cancer. Am J Obstet Gynecol. 2021 Feb;224(2):191.e1-191.e15. doi: 10.1016/j.ajog.2020.08.032. Epub 2020 Aug 15. PMID 32805208
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2008- September 2015. All recruitments were done in a medical clinic setting.
Pre-assignment Details: 69 participants enrolled, 12 participants did not participate on study (9) upgraded pathology, (2) screen failure and (1) withdrew.
Groups:
- Treatment: Single arm study, 52 mg levonorgestrel (Mirena) intrauterine device
Period: Overall Study
Arm/Group | Treatment
Started | 57
Completed | 47
Not Completed | 10
Not completed — Death | 2
Not completed — Unable to biopsy | 1
Not completed — Withdrawal by Subject | 4
Not completed — IUD expulsed | 1
Not completed — Lost to follow up | 2

BASELINE CHARACTERISTICS:
Groups:
- Levonorgestrel-releasing IUD: Single arm study, 52 mg levonorgestrel (Mirena) intrauterine device
Arm/Group | Levonorgestrel-releasing IUD
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45
  Black | 9
  Asian | 2
  Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 57
Body mass index (BMI) at diagnosis [Median (Full Range); unit: kg/m^2] | 45.5 [21 to 79]
Parity [Count of Participants; unit: Participants] — The number of times the participants gave birth.
  Participants
    Parous | 27
    Nonparous | 30
Menopausal status [Count of Participants; unit: Participants]
  Menopausal | 25
  Premenopausal | 32
Grade 1 Endometrioid Endometrial Cancer (G1EEC) [Count of Participants; unit: Participants] — Participants diagnosed with Grade 1 Endometrioid Endometrial Cancer (G1EEC). Population: Participants diagnosed with Grade 1 Endometrioid Endometrial Cancer (G1EEC).
  Participants
    Desires of future childbearing: number analyzed (Participants) | 49
    Desires of future childbearing | 3
    BMI of >40 kg/m2: number analyzed (Participants) | 49
    BMI of >40 kg/m2 | 5
    Multiple comorbidities: number analyzed (Participants) | 49
    Multiple comorbidities | 2
    Desires future childbearing +BMI of >40 kg/m2: number analyzed (Participants) | 49
    Desires future childbearing +BMI of >40 kg/m2 | 3
    BMI of >40 kg/m2 + multiple comorbidities: number analyzed (Participants) | 49
    BMI of >40 kg/m2 + multiple comorbidities | 6
    Desires future childbearing + BMI of >40 kg/ m2þmultiple comorbidities: number analyzed (Participants) | 49
    Desires future childbearing + BMI of >40 kg/ m2þmultiple comorbidities | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at 12 Month
Description: Will be defined as complete response or partial response based on the endometrial biopsy.
Time Frame: At 1 year
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
percentage of participants | 83 [72.7 to 90.3]

2. Primary Outcome: Efficacy of the Levonorgestrel Intrauterine Device (IUD)
Description: To determine the efficacy of the Levonorgestrel Intrauterine Device (IUD) to treat complex atypical hyperplasia (CAH) and grade 1 endometrioid endometrial carcinoma (G1 EEC), defined as complete regression disease. The primary efficacy endpoint was pathologic response rate (RR) at 12 months defined as complete response (CR) or partial response (PR). CR was defined as no evidence of cancer or hyperplasia with atypia in patients with (CAH) or EEC. PR was defined as CAH in patients with EEC. Progressive disease (PD) was defined as grade 2 endometrioid endometrial cancer or above in patients with EEC or the presence of any cancer in patients with CAH.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 47
Participants
  Complete Responders | 37
  Partial Responders | 2
  Stable Disease | 3
  Progressive Disease | 5

3. Secondary Outcome: Quality of Life Score Using the Short Form-36 (SF-36) Survey
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being (physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health); 2 summary scores (physical and mental component); and self evaluated change in health status (summary of health status). The score for subscale scores and 2 summary score is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Summary of health status is a 5-point Likert scale ranging from "0=much worse now" to "4=much better now". Higher subscale and summary score reflect better health status.
Time Frame: At baseline, 3 month, 6 month, 9 month and 12 month
Population: Number of participants analyzed differ for each row.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 57
score on a scale
  Physical Functioning Baseline: number analyzed (Participants) | 49
  Physical Functioning Baseline | 61.1 (31.2)
  Physical Functioning 3 month: number analyzed (Participants) | 46
  Physical Functioning 3 month | 65.0 (30.8)
  Physical Functioning 6 month: number analyzed (Participants) | 42
  Physical Functioning 6 month | 69.0 (29.6)
  Physical Functioning 9 month: number analyzed (Participants) | 40
  Physical Functioning 9 month | 68.3 (33.4)
  Physical Functioning 12 month: number analyzed (Participants) | 37
  Physical Functioning 12 month | 66.3 (31.9)
  Role-Physical Baseline: number analyzed (Participants) | 49
  Role-Physical Baseline | 55.1 (41.8)
  Role-Physical 3 month: number analyzed (Participants) | 47
  Role-Physical 3 month | 61.9 (38.8)
  Role-Physical 6 month: number analyzed (Participants) | 42
  Role-Physical 6 month | 69.0 (41.6)
  Role-Physical 9 month: number analyzed (Participants) | 40
  Role-Physical 9 month | 74.4 (38.2)
  Role-Physical 12 month: number analyzed (Participants) | 37
  Role-Physical 12 month | 74.3 (39.3)
  Role-Emotional Baseline: number analyzed (Participants) | 50
  Role-Emotional Baseline | 65.3 (40.9)
  Role-Emotional 3 month: number analyzed (Participants) | 46
  Role-Emotional 3 month | 61.6 (40.3)
  Role-Emotional 6 month: number analyzed (Participants) | 41
  Role-Emotional 6 month | 72.4 (37.2)
  Role-Emotional 9 month: number analyzed (Participants) | 40
  Role-Emotional 9 month | 71.7 (39.6)
  Role-Emotional 12 month: number analyzed (Participants) | 37
  Role-Emotional 12 month | 72.1 (40.5)
  Vitality Baseline: number analyzed (Participants) | 50
  Vitality Baseline | 50.0 (21.2)
  Vitality 3 month: number analyzed (Participants) | 46
  Vitality 3 month | 50.1 (25.0)
  Vitality 6 month: number analyzed (Participants) | 42
  Vitality 6 month | 57.5 (15.0)
  Vitality 9 month: number analyzed (Participants) | 40
  Vitality 9 month | 56.9 (21.5)
  Vitality 12 month: number analyzed (Participants) | 37
  Vitality 12 month | 51.9 (26.1)
  Mental health Baseline: number analyzed (Participants) | 50
  Mental health Baseline | 67.7 (21.7)
  Mental health 3 month: number analyzed (Participants) | 46
  Mental health 3 month | 67.7 (22.5)
  Mental health 6 month: number analyzed (Participants) | 42
  Mental health 6 month | 73.3 (18.0)
  Mental health 9 month: number analyzed (Participants) | 40
  Mental health 9 month | 73.1 (16.8)
  Mental health 12 month: number analyzed (Participants) | 37
  Mental health 12 month | 70.5 (21.4)
  Social functioning Baseline: number analyzed (Participants) | 50
  Social functioning Baseline | 68.5 (27.9)
  Social functioning 3 month: number analyzed (Participants) | 47
  Social functioning 3 month | 67.3 (29.9)
  Social functioning 6 month: number analyzed (Participants) | 42
  Social functioning 6 month | 77.7 (22.3)
  Social functioning 9 month: number analyzed (Participants) | 40
  Social functioning 9 month | 78.8 (26.1)
  Social functioning 12 month: number analyzed (Participants) | 37
  Social functioning 12 month | 72.0 (28.5)
  Pain Baseline: number analyzed (Participants) | 50
  Pain Baseline | 67.7 (25.3)
  Pain 3 month: number analyzed (Participants) | 47
  Pain 3 month | 70.5 (24.0)
  Pain 6 month: number analyzed (Participants) | 42
  Pain 6 month | 72.0 (24.3)
  Pain 9 month: number analyzed (Participants) | 40
  Pain 9 month | 73.5 (24.9)
  Pain 12 month: number analyzed (Participants) | 37
  Pain 12 month | 70.7 (23.4)
  General health Baseline: number analyzed (Participants) | 50
  General health Baseline | 55.6 (22.4)
  General health 3 month: number analyzed (Participants) | 47
  General health 3 month | 56.8 (22.2)
  General health 6 month: number analyzed (Participants) | 42
  General health 6 month | 60.8 (21.1)
  General health 9 month: number analyzed (Participants) | 40
  General health 9 month | 62.0 (20.0)
  General health 12 month: number analyzed (Participants) | 37
  General health 12 month | 60.1 (19.6)

ADVERSE EVENTS:
Time Frame: From baseline through 30 days following the IUD removal, up to 12 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 26/57
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=57)
Vaginal bleeding (Blood and lymphatic system disorders) | 26
Abdominal/Pelvic pain (Gastrointestinal disorders) | 9
Weight gain (Investigations) | 11
Breast pain (Reproductive system and breast disorders) | 3
Headache (Nervous system disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT00788671/Prot_SAP_000.pdf